CLINICAL TRIAL: NCT00551928
Title: A PHASE 3, MULTICENTRE, RANDOMIZED, CONTROLLED STUDY TO DETERMINE THE EFFICACY AND SAFETY OF LENALIDOMIDE, MELPHALAN AND PREDNISONE (MPR) Versus MELPHALAN (200 mg/m2) FOLLOWED BY STEM CELL TRANSPLANT IN NEWLY DIAGNOSED MULTIPLE MYELOMA SUBJECTS
Brief Title: Lenalidomide Melphalan and Prednisone Versus High Dose Melphalan in Newly Diagnosed Multiple Myeloma Patients
Acronym: MPRvsMEL200
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-209
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Newly Diagnosed Patients
Keywords: Multiple Myeloma; Lenalidomide; High dose Melphalan; Mobilization; CD34
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Lenalidomide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Oral therapy with Lenalidomide Melphalan and Prednisone.
  Interventions: Drug: Lenalidomide; Drug: Prednisone; Drug: Melphalan
- B (Active Comparator): High dose Melphalan therapy (200mg/sm)with autologous stem cell support, for 2 cycles every 4 months (only 1 cycle if the patient reached almost a VGPR after the 1st MEL200)
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — High dose Melphalan 200mg/sm with autologous stem cell support
  Arms: B
Drug: Lenalidomide — Six months of oral therapy with Lenalidomide 10mg/day given 21 days in every 28 days cycle with the combination ofMelphalan and steroids (day 22 to 28), for 6 cycles every 28 days.
  Arms: A
Drug: Prednisone — Given orally at the dose of 2 mg/Kg for 4 days followed by a 24 day rest period (days 5 to 28), for 6 cycles every 28 days
  Arms: A
Drug: Melphalan — Melphalan will be given orally at the dose of 0.18 mg/Kg for 4 days, followed by a 24 days rest period (day 5 to 28)for 6 cycles every 28 days
  Arms: A

SUMMARY:
To compare the efficacy of the combination of lenalidomide with low-dose melphalan versus high-dose melphalan in newly diagnosed, symptomatic MM patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient is 65 years old or younger at the time of signing the informed consent
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable double method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Negative serum β-human chorionic gonadotropin ( β-HCG) pregnancy test both 24 hours prior to beginning of therapy and then at 4 weeks intervals in women with regular menstrual cycles or every 2 weeks in women with irregular menstrual cycles during study treatment for subjects of childbearing potential
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of lenalidomide therapy.
* Patient was diagnosed with symptomatic multiple myeloma based on standard criteria (9), and has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours; measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan); bone marrow plasma cells>10%.
* Patient has a Karnofsky performance status ≥ 60%.
* Patient has a life-expectancy > 6 months
* Patient has not active infectious hepatitis type B or C, and has HIV negative test
* Patients must have an ejection fraction by ECHO or MUGA > 50% performed within 60 days prior to registration
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted. Patients unable to complete pulmonary function tests because of myeloma-related chest pain, must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):

  * Platelet count ≥ 75 x 109/L without transfusion support within 7 days before the test.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without the use of growth factors.
  * Corrected serum calcium ≤ 14 mg/dL (3.5 mmol/L).
  * Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal (ULN).
  * Alanine transaminase (ALT): ≤ 2.5 x the ULN.
  * Total bilirubin: ≤ 1.5 x the ULN.
  * Calculated or measured creatinine clearance: ≥ 30 mL/minute
* Patient has a baseline bone marrow sample available for cytogenetics, that will be processed and eventually centralized within each country.

Exclusion Criteria:

* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid; < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
* Pregnant or lactating females.
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
* Neuropathy of ≥ grade 2 severity.
* Patients previously diagnosed as bearing deep venous thrombosis or arterial thromboembolic event within the latest 12 months, or bearing a clear indication for anti-platelet or anticoagulant therapy or bearing a high risk of bleeding complications are ineligible for the sub-study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2007-06; Primary Completion 2022-06 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years

SECONDARY OUTCOMES:
Over all survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gay, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- Division of Hematology, AOU Città della Salute e della Scienza di Torino, Torino, Italy

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778
- [Derived] Cerrato C, Di Raimondo F, De Paoli L, Spada S, Patriarca F, Crippa C, Mina R, Guglielmelli T, Ben-Yehuda D, Oddolo D, Nozzoli C, Angelucci E, Cascavilla N, Rizzi R, Rocco S, Baldini L, Ponticelli E, Marcatti M, Cangialosi C, Caravita T, Benevolo G, Ria R, Nagler A, Musto P, Tacchetti P, Corradini P, Offidani M, Palumbo A, Petrucci MT, Boccadoro M, Gay F. Maintenance in myeloma patients achieving complete response after upfront therapy: a pooled analysis. J Cancer Res Clin Oncol. 2018 Jul;144(7):1357-1366. doi: 10.1007/s00432-018-2641-5. Epub 2018 Apr 19. PMID 29675792
- [Derived] Palumbo A, Cavallo F, Gay F, Di Raimondo F, Ben Yehuda D, Petrucci MT, Pezzatti S, Caravita T, Cerrato C, Ribakovsky E, Genuardi M, Cafro A, Marcatti M, Catalano L, Offidani M, Carella AM, Zamagni E, Patriarca F, Musto P, Evangelista A, Ciccone G, Omede P, Crippa C, Corradini P, Nagler A, Boccadoro M, Cavo M. Autologous transplantation and maintenance therapy in multiple myeloma. N Engl J Med. 2014 Sep 4;371(10):895-905. doi: 10.1056/NEJMoa1402888. PMID 25184862
- [Derived] Dunavin NC, Wei L, Elder P, Phillips GS, Benson DM Jr, Hofmeister CC, Penza S, Greenfield C, Rose KS, Rieser G, Merritt L, Ketcham J, Heerema N, Byrd JC, Devine SM, Efebera YA. Early versus delayed autologous stem cell transplant in patients receiving novel therapies for multiple myeloma. Leuk Lymphoma. 2013 Aug;54(8):1658-64. doi: 10.3109/10428194.2012.751528. Epub 2012 Dec 31. PMID 23194056
- [Derived] Larocca A, Cavallo F, Bringhen S, Di Raimondo F, Falanga A, Evangelista A, Cavalli M, Stanevsky A, Corradini P, Pezzatti S, Patriarca F, Cavo M, Peccatori J, Catalano L, Carella AM, Cafro AM, Siniscalchi A, Crippa C, Petrucci MT, Yehuda DB, Beggiato E, Di Toritto TC, Boccadoro M, Nagler A, Palumbo A. Aspirin or enoxaparin thromboprophylaxis for patients with newly diagnosed multiple myeloma treated with lenalidomide. Blood. 2012 Jan 26;119(4):933-9; quiz 1093. doi: 10.1182/blood-2011-03-344333. Epub 2011 Aug 11. PMID 21835953